CLINICAL TRIAL: NCT05629468
Title: Comparing Efficacy of Azithromycin and Probiotics for Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Mushayada Irshad, Prinicipal Investigator, Pak Emirates Military Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A/28/EC/337/2021
Record Dates: First submitted 2022-11-09; First posted 2022-11-29 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Azithromycin; Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azithromycin and Topical (Active Comparator): group A (n=25) received tab. azithromycin 250mg oral on alternate days and topical cream benzoyl peroxide 4% twice a day daily for a period of 3 months
  Interventions: Drug: Azithromycin; Drug: Benzoyl Peroxide 4 % Topical Cream
- Probiotics and Topical (Experimental): group B (n=25) received Probiotic sachet oral once a day everyday and topical cream benzoyl peroxide 4% twice a day daily for a period of 3 months
  Interventions: Drug: Probiotic Formula; Drug: Benzoyl Peroxide 4 % Topical Cream
- Azithromycin and Probiotics and Topical (Other): combination group C (n=25) received tab. azithromycin 250mg oral on alternate days, Probiotic sachet oral once a day everyday and topical cream benzoyl peroxide 4% twice a day daily for a period of 3 months
  Interventions: Drug: Azithromycin; Drug: Probiotic Formula; Drug: Benzoyl Peroxide 4 % Topical Cream

INTERVENTIONS:
Drug: Azithromycin — antibiotic
  Other Names: "Zetro" by "Getz Pharma"
  Arms: Azithromycin and Probiotics and Topical; Azithromycin and Topical
Drug: Probiotic Formula — probiotics
  Other Names: "Hi-Flora" by "Unicare Bioceuticals"
  Arms: Azithromycin and Probiotics and Topical; Probiotics and Topical
Drug: Benzoyl Peroxide 4 % Topical Cream — topical cream
  Other Names: "Benoxyl" by "Glitz pharma"

SUMMARY:
the goal of this clinical trial is to measure the efficacy of probiotics for treatment of acne vulgaris, to compare it with azithromycin and to measure the synergistic effect of azithromycin and probiotics for treatment of acne vulgaris

DETAILED DESCRIPTION:
this study aims to answer this research question: in patients of acne vulgaris, is use of probiotics as efficacious as azithromycin in treating acne lesions & improving quality of life? total 75 patients were divided into 3 groups. group A received azithromycin, group B received probiotics and group C received both drugs. a topical cream was also advised to all groups. outcome was measured as reduction in total lesion count and improvement in patients' quality of life via reduction in Dermatology Life Quality Index score.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Patients of Mild and Moderate acne
* Aged between 15 and 35 years

Exclusion Criteria:

* Severe acne or any systemic inflammatory disease
* Other oral treatment for acne
* Allergic to any drug being used in the study
* Pregnancy
* PCOs
* Any drug which can interact with azithromycin

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
change or reduction in the Total Lesion Count | at start of the study (baseline), 2 weeks (1st follow up visit), 4 weeks (2nd follow up visit), 8 weeks (3rd follow up visit) and 12 weeks (4th follow up visit).
  number of acne lesions are counted at every follow up to see whether lesions are reduced than the baseline or not

SECONDARY OUTCOMES:
change or reduction in the Dermatology Life Quality Index score | at start of the study (baseline) and 12 weeks (last follow up visit).
  improvement in patients' quality of life was assessed to see whether the score has been reduced than the baseline score or not. it was assessed by a 10-item self assessment questionnaire i.e Dermatology Life Quality Index. the score ranges between 0 to 30. higher score means worst outcome and the lower score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Akbar W Syed, PhD, Study Director — Riphah International University, Islamabad
Locations (1):
- PEMH, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No